CLINICAL TRIAL: NCT04702399
Title: Hyaluronic Acid for the Prevention of Endocavitary Synechiae After Myomectomy by the Abdominal Route: Prospective,Randomized, Multicenter and Pilot Study.
Brief Title: Hyaluronic Acid for the Prevention of Endocavitary Synechiae After Myomectomy
Acronym: PREVENDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP200247
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-11

CONDITIONS: Patients With an Indication for Myomectomy or Polymyomectomy
Keywords: Synechia; Myomas; Myomectomy; Polymyomectomy; Gynaecology
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEL GROUP (Experimental): Intracavitary application of an anti-adhesion hyaluronic acid gel (HYALOBARRIER® GEL ENDO)
  Interventions: Device: GEL GROUP
- CONTROL GROUP (No Intervention): No Intervention

INTERVENTIONS:
Device: GEL GROUP — Application of an anti-adhesion gel (HYALOBARRIER® GEL ENDO) in the uterine cavity
  Arms: GEL GROUP

SUMMARY:
PREVENDO is a prospective, multicenter, pilot, and randomized study in 2 parallel arms and single blind, evaluating the proportion of endometrial synechiae 6 weeks after surgery in patients undergoing abdominal myomectomy or polymyomectomy, according to the application or not of an anti-adhesion gel (HYALOBARRIER® GEL ENDO)

DETAILED DESCRIPTION:
Myomas are a common pathology affecting a large population of women of reproductive age. Depending on their location and the patient's symptoms, surgical removal of fibroids may be indicated.

Interstitial or subserous myomas are accessible through the abdominal route (laparotomy or minimally invasive surgery).

The impact of this surgery on the endometrial cavity and the risk of post-surgery synechiae is poorly understood, although it is essential, especially in a population of women wishing to preserve their fertility. In order to reduce and prevent endometrial synechia formation, we suggest PREVENDO study which consist in the systematic intracavitary placement of an anti-adhesion gel (HYALOBARRIER® GEL ENDO) immediately after surgery in patients undergoing abdominal myomectomy or polymyomectomy (laparotomy, laparoscopy, robot-assisted laparoscopy) and the evaluation of the proportion of endometrial synechiae 6 weeks after surgery in patients during diagnostic hysteroscopy performed 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Of childbearing age
3. Indication of myomectomy / polymyomectomy by laparotomy / laparoscopy / robot-assisted laparoscopy
4. FIGO 2 to 6 classification myomas

Exclusion Criteria:

1. History of intra uterine synechia treatment
2. Uterine malformation
3. Patients under legal protection measure (guardianship or curatorship) or under security measure
4. Pregnant or breastfeeding women
5. Absence of health insurance; or patient with AME
6. Absence of free, informed and written consent
7. Endometrial synechia before operation (grade 1-3) (assessed by systematic diagnostic hysteroscopy)
8. Patient with upper genital infection
9. Hypersensibility to hyaluronic acid

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with endometrial synechiae | 6 weeks after surgery (+/-2weeks)
  The evaluation of the proportion of endometrial synechiae in patients udergoing abdominal myomectomy or polymyoomectomy, during diagnostic hysteroscopy performed 6 weeks after surgery.

SECONDARY OUTCOMES:
Proportion of patients with moderate or severe endometrial synechiae | 6 weeks after surgery (+/-2 weeks)
  The evaluation of the proportion of endometrial synechiae in patients udergoing abdominal myomectomy or polymyoomectomy, during diagnostic hysteroscopy performed 6 weeks after surgery.Severity is assessed using the American Fertility Society score (AFS)
Proportion of patients with increased of menstrual bleeding or menstrual bleeding time | 6 weeks after surgery (+/- 2 weeks)
  Assessed subjectively by patients (Increase vs No increase)
The quality of life | 6 weeks after surgery (+/- 2 weeks)
  Assessed using EQ-5D-5L questionnary. The EQ5D uses a Likert scale which assesses five states (mobility, self care, usual care, pain and discomfort and anxiety and depression) at five different levels - none, slight, moderate, severe or unable to perform. Levels are coded 1-5 and a total score is then generated.
Dysmenorrhea | 6 weeks after surgery (+/- 2 weeks)
  Assessed using the visual analogic scale (VAS)
Spontaneous pelvic pain | 6 weeks after surgery (+/- 2 weeks)
  Assessed using the visual analogic scale (VAS)
Metrorragia | 6 weeks after surgery (+/- 2 weeks)
  Assessed subjectively by patients

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy Doctor CANLORBE, Study Director — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.